CLINICAL TRIAL: NCT03660371
Title: Internal Limiting Membrane Peeling in Proliferative Diabetic Retinopathy Patients Undergoing Vitrectomy for Vitreous Hemorrhaging
Brief Title: ILM Peeling in PDR Patients Undergoing PPV for VH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush Eye Associates (Other)
Responsible Party: Principal Investigator, Sloan W. Rush, MD, Physician, Rush Eye Associates
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Retina 2
Record Dates: First submitted 2018-09-04; First posted 2018-09-06 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2021-11

CONDITIONS: Diabetic Retinopathy; Macular Edema
MeSH Terms: conditions — Diabetic Retinopathy; Macular Edema | interventions — Predictive Value of Tests

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PPV/MP (Experimental): Study Group: Subjects undergo internal limiting membrane (ILM) peeling during vitrectomy for the indication of diabetic vitreous hemorrhaging
  Interventions: Procedure: PPV/MP
- PPV without MP (Active Comparator): Control Group: Subjects do not undergo ILM peeling during vitrectomy for the indication of diabetic vitreous hemorrhaging
  Interventions: Procedure: PPV without MP

INTERVENTIONS:
Procedure: PPV/MP — Internal limiting membrane (ILM) peeling during vitrectomy for the indication of diabetic vitreous hemorrhaging
  Arms: PPV/MP
Procedure: PPV without MP — No internal limiting membrane (ILM) peeling during vitrectomy for the indication of diabetic vitreous hemorrhaging
  Arms: PPV without MP

SUMMARY:
Subjects undergoing ILM peeling during vitrectomy will have better visual acuity and lower rates of DME to control subjects

DETAILED DESCRIPTION:
Proliferative diabetic retinopathy (PDR) and diabetic macular edema (DME) frequently occur together in patients with diabetic retinopathy In the landmark study Protocol S, about 30% of PDR subjects had DME at baseline and 53% of subjects receiving panretinal photocoagulation (PRP) underwent treatment for DME during the 2-year study interval. Vitreous hemorrhaging is one of the most common indications for pars plana vitrectomy (PPV) in patients with PDR. PDR patients undergoing PPV for the treatment of vitreous hemorrhaging often have coexisting DME, although it is often difficult to identify preoperatively because of the media opacification from the vitreous hemorrhage. Following successful PPV and vitreous hemorrhage resolution, PDR patients may then require prolonged DME treatment with repetitive intravitreal injections and/or focal lasers.

PPV with internal limiting membrane (ILM) peeling has been reported to reduce retinal edema and improve visual acuity in patients with DME. Although numerous studies report favorable outcomes in patients undergoing PPV with ILM peeling for the surgical indication of DME, there are presently not any studies evaluating ILM peeling in PDR patients undergoing PPV for the primary indication of vitreous hemorrhaging. Performing ILM peeling in conjunction with the usual techniques for addressing a vitreous hemorrhage (i.e. endolaser PRP, endodiathermy, etc.) during PPV may offer the benefits of better postoperative visual acuity and/or fewer postoperative treatments required to manage DME. In this randomized controlled trial, the authors evaluate the merits of ILM peeling in PDR patients undergoing PPV for the primary indication of vitreous hemorrhaging.

ELIGIBILITY:
Inclusion Criteria:

1. Subject age is 18-85 years.
2. Subject consents to study participation and is capable of 6 months of follow-up.
3. The subject has type I or II Diabetes Mellitus with active PDR in the study eye.
4. Best-corrected spectacle visual acuity (BCSVA) on the Snellen eye chart ranges from 20/40 to hand motions in the study eye.
5. The subject is determined to need a PPV for the indication of reduced BCSVA from vitreous hemorrhaging without substantial vitreoretinal (VR) adhesion (Grades 0 and 1).

Exclusion Criteria:

1. Subject is known to have a significant retinal/optic nerve disease otherwise unrelated to Diabetes Mellitus, which in the opinion of the examiner is responsible for two or more lines of reduced BCSVA (macular degeneration, optic neuritis, glaucoma, amblyopia, etc.) in the study eye.
2. Subject is known to have macular ischemia, which in the opinion of the examiner, is responsible for two or more lines of reduced BCSVA in the study eye.
3. Subject has a significant corneal opacity, which in the opinion of the examiner, is responsible for two or more lines of reduced BCSVA (corneal scar, ectasia, etc.) in the study eye.
4. Subject has a retinal detachment in the study eye.
5. Subject has had a previous vitrectomy (anterior or PPV) in the study eye.
6. Subject has uncontrolled neovascular glaucoma (intraocular pressure > 30 mmHg despite medical/surgical treatment) in the study eye.
7. Subject has uncontrolled hypertension (systolic > 200 mmHg or diastolic > 120 mmHg) despite adherence to a multiple anti-hypertensive medication regimen.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2018-09-04 (Actual); Primary Completion 2020-03-04 (Actual); Study Completion 2020-03-04 (Actual)

PRIMARY OUTCOMES:
BCVA | 6 months
  best-corrected visual acuity

CONTACTS AND LOCATIONS:
Overall Officials: Sloan Rush, Study Chair — panhandle eye group
Locations (1):
- Hospital La Carlota, Montemorelos, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: No